CLINICAL TRIAL: NCT01909518
Title: Detection of Early Esophageal Squamous Neoplasia by Using Virtual Chromoendoscopy and Probe-based Confocal Laser Endomicroscopy
Brief Title: Detection of Early Esophageal Squamous Neoplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2013SDU-QILU-G02
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Esophageal Squamous Intraepithelial Neoplasia
Keywords: Esophageal Squamous Intraepithelial Neoplasia; surface maturation scoring; probe-based confocal laser endomicroscopy; virtual chromoendoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — endoscopic biopsies will be taken at suspicious lesions
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pCLE examination: pCLE is used to distinguish the suspected lesions detected by I-SCAN in esophagus

SUMMARY:
The aim of the present study：

1. To investigate the diagnosing value of pCLE for early esophageal squamous neoplasia.
2. To assess the detection rate of early esophageal squamous neoplasia by virtual chromoendoscopy

DETAILED DESCRIPTION:
Probe-based confocal laser endomicroscopy (pCLE; Cellvizio, Mauna Kea Technologies, Paris, France) is a newly developed endoscopic device and has shown its value for diagnosing Barrett's esophagus, colonal polyps and etc. However, none research has focus on early esophageal squamous neoplasia until now. Previous diagnosis of early esophageal neoplasia is based on the lugol staining which is time wasting and have many adverse events.Other researches have suggested virtual chromoendoscopys are beneficial for screening esophageal tumors. Therefore, the aim of the present study is 1.To investigate the diagnosing value of pCLE for early esophageal squamous neoplasia according to the surface maturation scoring(SMS) diagnostic criteria and 2. To assess the detection rate of early esophageal squamous neoplasia by virtual chromoendoscopy(I-SCAN).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 50 and 80 years old
* Patients undergo screening endoscopy or histologically verified esophageal squamous intraepithelial neoplasia before.

Exclusion Criteria:

* Advanced esophageal, gastric or duodenal cancer
* History of upper GI tract surgery
* Coagulopathy or acute GI bleeding
* Pregnant or breast-feeding (for females)
* Impaired renal function
* Allergy to fluorescein sodium
* Inability to provide informed consent.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of pCLE on early esophageal squamous neoplasia | 6 month
  Patients will be prospectively recruited to evaluate the diagnostic sensitivity, specificity and accuracy of early esophageal squamous neoplasia by using probe-based confocal laser endomicroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD. PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China